CLINICAL TRIAL: NCT01116713
Title: Preoperative Dexamethasone Reduces Postoperative Pain, Nausea and Vomiting Following Mastectomy for Breast Cancer.
Brief Title: Effect of Dexamethasone in Postoperative Symptoms After Mastectomy for Breast Cancer
Acronym: dxt2010brca
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Alejandro Gonzalez-Ojeda, Mexican Institute of Social Security
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Dxt-2010-breast cancer
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2010-05-05 (Estimated); Status verified 2010-05

CONDITIONS: Postoperative Pain; Postoperative Nausea; Postoperative Vomiting
Keywords: Mastectomy; Breast cancer; Postoperative pain; Postoperative nausea and vomiting
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone group (Active Comparator): This group of patients received intravenous dexamethasone (8 mg) 60 minutes before skin incision.
  Interventions: Drug: intravenous dexamethasone
- Placebo group (Placebo Comparator): Patients of these group received homologated placebo 60 minutes before skin incision.
  Interventions: Drug: Homologated placebo.

INTERVENTIONS:
Drug: intravenous dexamethasone — One dose of intravenous dexamethasone (8 mg) 60 minutes before skin incision.
  Other Names: no other intervention
  Arms: Dexamethasone group
Drug: Homologated placebo. — Patients of the control group received homologated placebo 60 minutes before skin incision
  Other Names: no other intervention
  Arms: Placebo group

SUMMARY:
Postoperative pain, nausea and vomiting (PONV) are the most common complications after anesthesia and surgery. Women undergoing mastectomy with axillary dissection are at a particularly high risk for the development of PONV and an incidence of 60-80% in patients receiving no antiemetic has been reported. Emetic episodes predispose to aspiration of gastric contents, wound dehiscence, psychological distress, and delayed recovery and discharge times. These justify the use of prophylactic antiemetics in women scheduled for mastectomy. Most of the currently used antiemetics, including antihistamines, butyrophenones and dopamine receptor antagonists have been reported to cause occasional undesirable adverse effects, such as excessive sedation, hypotension, dry mouth, dysphoria, hallucinations and extrapyramidal signs. Antiserotonins (e.g., ondansetron) are available for the prevention and treatment of PONV in patients undergoing various types of surgery [4]. However, the use of prophylactic antiemetic therapy with antiserotonins has been criticized for being too expensive.

Dexamethasone was first reported to be an effective antiemetic regimen in patients receiving cancer chemotherapy.

The purpose of this study was to evaluate the efficacy of dexamethasone treatment for reducing pain and PONV as well as analgesic and antiemetic requirements in women undergoing general anesthesia for mastectomy with axillary lymph node dissection.

DETAILED DESCRIPTION:
Breast cancer is the most frequent malignant neoplasm worldwide. In emerging countries such as Mexico, there has been an increase in its frequency and mortality [1, 2] and it is the second most frequent neoplasm after cervical carcinoma. Between 25,000 and 30,000 new cases are diagnosed annually. Unfortunately, only a few women have regular mammography screening so the proportion of patients with locally advanced disease at diagnosis is high. In 2003, only 5-10% of newly diagnosed cases in Mexico were clinical stages 0 or I [2]. Surgical resection with axillary lymph node dissection constitutes the treatment of choice associated with neoadjuvant therapy and postoperative chemotherapy and/or radiation therapy.

Postoperative pain, nausea and vomiting (PONV) are the most common complications after anesthesia and surgery. Women undergoing mastectomy with axillary dissection are at a particularly high risk for the development of PONV and an incidence of 60-80% in patients receiving no antiemetic has been reported. Emetic episodes predispose to aspiration of gastric contents, wound dehiscence, psychological distress, and delayed recovery and discharge times. These justify the use of prophylactic antiemetics in women scheduled for mastectomy. Most of the currently used antiemetics, including antihistamines, butyrophenones and dopamine receptor antagonists have been reported to cause occasional undesirable adverse effects, such as excessive sedation, hypotension, dry mouth, dysphoria, hallucinations and extrapyramidal signs. Antiserotonins (e.g., ondansetron) are available for the prevention and treatment of PONV in patients undergoing various types of surgery. However, the use of prophylactic antiemetic therapy with antiserotonins has been criticized for being too expensive.

Dexamethasone was first reported to be an effective antiemetic regimen in patients receiving cancer chemotherapy. Some authors have reviewed the available randomized trials (1996-2001) regarding perioperative single-dose steroid administration and found that dexamethasone had antiemetic and analgesic effects in various types of operations. One ot this studies demostrated that intravenous dexamethasone at 4 mg was effective for the prevention of PONV following breast surgery but they could not demonstrate any difference in postoperative pain.

The purpose of this study was to evaluate the efficacy of dexamethasone treatment for reducing pain and PONV as well as analgesic and antiemetic requirements in women undergoing general anesthesia for mastectomy with axillary node dissection.

Patients and Methods Patients Between June and August 2009, 70 patients undergoing mastectomy with axillary dissection were studied in a prospective, randomized, double-blind clinical trial. Patients were randomized to receive intravenous dexamethasone (8 mg) or homologated placebo 60 minutes before skin incision, using an equal number of blinded envelopes. Patients of American Society of Anesthesiologists classes III and IV were excluded. Further exclusion criteria were age more than 80 years; pregnancy; active menstruation; treatment with steroids; severe diabetes mellitus (serum HbA1c > 8%); use of opioids, sedatives or any kind of analgesics less than one week before mastectomy, or a history of alcohol or drug abuse. Patients with any history of motion sickness and ⁄or previous PONV after any surgical procedure were excluded. All patients were admitted to the hospital one day before the operation and were followed from hospital admission until 30 days after the surgical procedure to detect any medical or surgical morbidity.

Anesthesia and surgery All patients underwent a standardized general anesthesia procedure and none of them received any preanesthetic medication. Induction used intravenous propofol (2 mg/kg body weight) and fentanyl (3-5 mcg/kg). Vecuronium bromide (0.1 mg/kg) was used to facilitate tracheal intubation. Anesthesia was maintained with 2-3% sevoflurane and 66% nitrous oxide in oxygen. Ventilation was controlled mechanically and maintained constant throughout surgery using an anesthetic and respiratory gas analyzer for monitoring.

All patients were monitored with indirect determinations of arterial pressure and heart rate using standard techniques, as well as the expired CO2 content and oxygen blood saturation. Afterwards, all patients were extubated and transferred to the immediate postsurgical care unit with cardiovascular and oxygen monitoring.

Surgical procedures All patients were treated according to the preoperative clinical stage with radical mastectomy or breast conservative surgery with lymph node axillary dissection by the same surgical team. In all patients, closed suction drains were placed in the region subjected to surgery and were removed during the following days. Chemotherapy and/or radiotherapy were administered 3-4 weeks after uncomplicated surgical resections.

Analgesia and antiemetic therapies Pain was assessed immediately on return to the recovery room and at 6, 12 and 24 h after the operation using a visual analogue scale (VAS; 0 = no pain to 10 = most severe pain). Analgesia was given as intravenous sodium ketorolac (30 mg every 8 hours) and intravenous tramadol infusion (50 mg) was used as a backup analgesic medication. The incidence of PONV was recorded immediately on return to the recovery room and at 6, 12 and 24 h after the operation, using a three point ordinal scale (0 = none, 1 = nausea, 2 = retching, 3 = vomiting). Nausea was defined as a subjectively unpleasant sensation associated with awareness of the urge to vomit, retching was defined as the labored, spasmodic, rhythmic contraction of the respiratory muscles without the expulsion of gastric contents, and vomiting was defined as the forceful expulsion of gastric contents from the mouth. Intravenous ondansetron (4-8 mg) was given for antiemetic treatment on demand.

Data collection and statistical analysis Postoperative complications were recorded during hospitalization and the patients were followed up to 30 days after discharge. Additional data collected included patient age, body mass index (BMI), any history of smoking and neoadjuvant chemotherapy, anesthesia and operation time and the frequency of use of analgesic and antiemetic drugs. These parameters were summed and compared between the dexamethasone and placebo groups.The study endpoints were postoperative nausea and vomiting, and pain measured by the VAS and the need for additional analgesic and antiemetic drugs.

The sample size was predetermined. We expected a 35% difference in the incidence of nausea and vomiting between groups. The alpha error was set at 0.05 and beta error at 0.20; n = 35 patients for each group was considered adequate, according to a power analysis. Results are expressed as percentages and as the mean ± standard deviation (SD). Student's t test, the Chi-squared test or Fisher's Exact Test were used for the analysis of quantitative and qualitative data, respectively. Differences were considered statistically significant at p < 0.05.

Ethical considerations The study was conducted according to the principles of the Declaration of Helsinki of 1989 and the Mexican Health Guidelines. The Ethical and Research Committees of the Oncologic Institute, approved all protocols. Full, written informed consent was obtained from all patients before their inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classes I-II female patients with breast cancer scheduled for surgical treatment; mastectomy plus axillary node dissection.

Exclusion Criteria:

* American Society of Anesthesiologists classes III and IV.
* Age more than 80 years; pregnancy; active menstruation; treatment with steroids; severe diabetes mellitus (serum HbA1c > 8%); use of opioids, sedatives or any kind of analgesics less than one week before mastectomy, or a history of alcohol or drug abuse.
* Patients with any history of motion sickness and or previous postoperative nausea and vomiting after any surgical procedure.

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Pain was assessed immediately on return to the recovery room and at 6, 12 and 24 h after the operation using a visual analogue scale (VAS; 0 = no pain to 10 = most severe pain). | 24 hours
  The pain intensity was recorded by a member of the team, blinded to the interventional manouver. A visual analogue scale for pain was used. The patient stablished the pain intensity and the researcher captured el number level. The information was obtained in the recovery room after the patient was monitorized and blood pressure and oxigen blood content values were normal. The information was obtained after 6, 12 and 24 hours after the surgical procedure.

SECONDARY OUTCOMES:
The incidence of nausea and vomiting was recorded immediately on return to the recovery room and at 6, 12 and 24 h after the operation, using a three point ordinal scale (0 = none, 1 = nausea, 2 = retching, 3 = vomiting). | 24 hours
  The presence of nausea and vomiting was recorded by a member of the team, blinded to the interventional manouver. A visual analogue scale for pain was used. The information was classified as asymptomatic (0), presence of nausea (1), retching (2) and vomiting (3) . The information was obtained in the recovery room after the patient was monitorized and blood pressure and oxigen blood content values were normal. The information was obtained after 6, 12 and 24 hours after the surgical procedure.
Total dose of backup analgesic and antiemetic medication administrated to each patient | 24 hours
  Total dose of backup analgesic and antiemetic medication were recorded during the first 24 hours after the surgical procedure.
Morbidity and mortality after mastectomy | 30 days
  Evaluation of any surgical or medical complication after surgery as well as mortalitiy 30 days after surgical treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Gonzalez-Ojeda, M.D., Ph.D., Study Director — Instituto Mexicano del Seguro Social
Locations (2):
- Mexico (2):
  - Breast Clinic. Oncologic Institute of Jalisco, Guadalajara, Jalisco
  - Research Unit in Clinical Epidemiology, Specialties Hospital. Mexican Institute of Sociaql Security, Guadalajara, Jalisco

REFERENCES:
- [Derived] Gomez-Hernandez J, Orozco-Alatorre AL, Dominguez-Contreras M, Oceguera-Villanueva A, Gomez-Romo S, Alvarez Villasenor AS, Fuentes-Orozco C, Gonzalez-Ojeda A. Preoperative dexamethasone reduces postoperative pain, nausea and vomiting following mastectomy for breast cancer. BMC Cancer. 2010 Dec 23;10:692. doi: 10.1186/1471-2407-10-692. PMID 21182781